CLINICAL TRIAL: NCT06852625
Title: Autologous Tolerogenic Dendritic Cells (ATDC) for Highly Sensitized Kidney Transplant Recipients
Acronym: ATDC-PICI
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-519978-39-00
Record Dates: First submitted 2025-02-14; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): An algorithm has been designed to rank highly sensitized patients on the waiting list for kidney transplantation according to their likelihood of obtaining a suitable donor within the upcoming 12 months. The algorithm was designed based on an analysis of an immunologically matched historical cohort using data from the OCATT registry.
  Patients will be selected in accordance with the algorithm and proposed for inclusion in the study in a sequential manner until the required number of patients has been reached (n=30). Given the unpredictability and reduced likelihood of obtaining a compatible deceased kidney donor within an acceptable time frame for this study, the total number of patients to be included will be 2x superior to those who will receive treatment with ATDC (n=15).
  * 30 highly sensitized patients will be pre-included in the study.
  * The first 15 highly sensitized patients that obtain a compatible deceased kidney donor will receive study treatment.
  Interventions: Biological: Autologous Tolerogenic Dendritic Cells

INTERVENTIONS:
Biological: Autologous Tolerogenic Dendritic Cells — • Autologous Tolerogenic Dendritic Cells (D+1 to D+3 post-transplantation), ATDC, 1 million ATDC/Kg over a period of 30 minutes (up to 1 hour) will administer between Day 1 and Day 3 after transplantation.

SUMMARY:
The ATDC-PICI study is a Phase Ib, single-arm, prospective, non-randomized, multicentric trial, to evaluate the safety of ATDC cell product as adjunctive therapy to standard of care (SOC) in highly sensitized kidney transplant recipients.

DETAILED DESCRIPTION:
The study population is sensitized kidney transplant candidates (cPRA ≥ 90%) between 18 and 65 years.

An algorithm has been designed to rank highly sensitized patients on the waiting list for kidney transplantation according to their likelihood of obtaining a suitable donor within the upcoming 12 months. The algorithm was designed based on an analysis of an immunologically matched historical cohort using data from the OCATT registry.

Patients will be selected in accordance with the algorithm and proposed for inclusion in the study in a sequential manner until the required number of patients has been reached (n=30). Given the unpredictability and reduced likelihood of obtaining a compatible deceased kidney donor within an acceptable time frame for this study, the total number of patients to be included will be 2x superior to those who will receive treatment with ATDC (n=15).

* 30 highly sensitized patients will be pre-included in the study.
* The first 15 highly sensitized patients that obtain a compatible deceased kidney donor will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Highly sensitized (cPRA ≥ 90%) kidney transplant candidates between 18 and 65 years old.
2. To be selected by the algorithm according to probability of kidney transplantation in the upcoming 12months.
3. Adequate venous access and absence of contraindications for leukoapheresis.
4. Women of childbearing age must take contraceptive measures.
5. Must have given written informed consent

Exclusion Criteria:

1. Subjects with active TB.
2. Patients on the waiting list multiple organ transplants.
3. A significantly abnormal general serum screening lab result defined as WBC<3.0x103/ml, Hgb<8.0 g/dL, platelet count <100x103/ml, SGOT>3x upper limit.
4. HIV-positive subjects.
5. Subjects who test positive for HBV infection [positive HBVsAg or HBVeAg/DNA] or HCV infection [RNA+].
6. Subjects with active CMV or EBV infection as defined by positive PCR.
7. Subjects with a known history of previous myocardial infarction within one year of screening.
8. Subjects with a history of clinically significant thrombotic episodes, and subjects with active peripheral vascular disease.
9. Patients with a kidney disease with high risk of recurrence and/or complement-associated kidney disease (aHUS, etc).
10. Pregnant and lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Side effects of ATDC cell product in highly sensitized patients who received a kidney from a deceased donor. | at day 1 and day 3
  Proportion of patients with toxicity/side effects during and after administration.

SECONDARY OUTCOMES:
Rate of infectious disease that required hospitalization at 6 and 12 months. | at 6 months and 12 months.
  Proportion of patients with severe or serious infections at 6 months and 12 months.
To evaluate incidence of biopsy proven acute rejection episodes in patients treated with ATDC as adjunctive therapy to SOC | at 3 and 12months after transplantation.
  Incidence of BPAR at 3 and 12months after transplantation.
To evaluate renal function up to 1 year after transplantation | at 3, 6 and 12 months after transplantation
  Renal function at 3, 6 and 12 months after transplantation as assessed by estimated glomerular filtration rate (eGFR)
To evaluate renal function up to 1 year after transplantation | at 3, 6 and 12 months after transplantation
  Renal function at 3, 6 and 12 months after transplantation as assessed by serum/plasma creatinine levels
To evaluate patient survival | at 12 months after transplantation
  Patient survival at 12 months after transplantation
To evaluate graft survival | at 12 months after transplantation
  Graft survival at 12 months after transplantation
To characterize the immunophenotype status. | 24 months
  Define the different cell subtypes in circulating cells, as well as the functionality of T and B cells using ELISpot and Fluorospot techniques

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Fundació Puigvert, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic Barcelona, Barcelona, Barcelona
  - Hospital Universitari Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No